CLINICAL TRIAL: NCT04788693
Title: Effects of Gait Rehabilitation With Motor Imagery in People With Parkinson's Disease
Acronym: GAITimagery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Asociación Parkinson Valencia (Other)
Responsible Party: Principal Investigator, Constanza San Martín, Associate Lecturer professor at the Department of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1557673
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
Keywords: Gait rehabilitation; Motor imagery; Biomechanics of gait; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: To ensure masking, the raters physiotherapist, and data analysis researcher, will be blinded to the participant's allocation. Although participants and treating physiotherapists cannot be totally blinded to the intervention performed, the hypothesis and objectives of the study will be hidden from them. At the same time, all participants will be instructed not to disclose information regarding their intervention to the raters' physiotherapists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor imagery and gait training group (Experimental): Gait training twice a week for six weeks. Each rehabilitation session is composed of an initial 5 minutes of warm-up exercises (general mobility, coordination, strength, flexibility, balance, and breathing), followed by 45 minutes of gait training with motor imagery exercises and a final 10 minutes of muscle stretching.
  In the central 45 minutes of the session, exercises will be developed to improve objective characteristics of the gait-related to spatiotemporal and kinematic parameters. Objective and subjective feedback will be used for each exercise (cues). In an interspersed way, motor imagery exercises will be carried out where participants must rehearse or simulate mentally each gait exercise that will be developed in the session.
  Interventions: Other: Physical rehabilitation of gait with motor imagery
- Gait training group without motor imagery (Active Comparator): Gait training twice a week for six weeks. Each rehabilitation session is composed of an initial 5 minutes of warm-up exercises (general mobility, coordination, strength, flexibility, balance, and breathing), followed by 45 minutes of gait training with motor imagery exercises and a final 10 minutes of muscle stretching.
  In the central 45 minutes of the session, exercises will be developed to improve objective characteristics of the gait-related to spatiotemporal and kinematic parameters. Objective and subjective feedback will be used for each exercise (cues). In the periods that the experimental group performs the motor imagery exercises, the control group will take breaks.
  Interventions: Other: Physical rehabilitation of gait without motor imagery

INTERVENTIONS:
Other: Physical rehabilitation of gait with motor imagery — Physical rehabilitation of gait is a type of non-invasive treatment that seeks to change the way of performing a task or motor function (in this case, gait) through movement modification and corrected repeated practice, taking into account the alterations, limitations and considerations related to the disease suffered by the person. In this intervention, in addition to physical exercise to correct gait, mental exercises will be included in which the patient visualizes himself performing the exercises that he will then develop with the body.
  Other Names: GAITimagery program
  Arms: Motor imagery and gait training group
Other: Physical rehabilitation of gait without motor imagery — Physical rehabilitation of gait is a type of non-invasive treatment that seeks to change the way of performing a task or motor function (in this case, gait) through movement modification and corrected repeated practice, taking into account the alterations, limitations and considerations related to the disease suffered by the person. Motor imagery exercises are not included in this program.
  Other Names: Gait physiotherapy program
  Arms: Gait training group without motor imagery

SUMMARY:
This study aims to determine whether gait physiotherapy combined with motor imagery exercises has a superior effect than gait physiotherapy without motor imagery in people with Parkinson's disease. To do this, a six-week training program will be carried out twice a week, where walking exercises and motor imaging will be performed in the experimental group while walking exercises only, will be conducted in the control group. Motor imagery exercises consist of developing a mental exercise by which an individual rehearses or simulates a given action. We hypothesize that participants who perform motor imagery exercises have better results than participants who train without imagery exercises. To analyze the effect of the programs will be assess the gait, the functionality in activities of daily living, the motor capacity, and the perception of the quality of life of the participants.

DETAILED DESCRIPTION:
Background:

Motor imagery (MI) is a novel technique in neurorehabilitation. Current evidence supports the ability of people diagnosed with Parkinson's disease (PD) to carry out this technique. However, the trials that assess its effectiveness in this pathology are scarce. In some physical rehabilitation programs, MI is introduced to conventional treatment or, MI can be combined with observation of images or neurofeedback. At present, the effect of this technique has been studied in highly heterogeneous variables, including both motor and cognitive abilities or performance of activities of daily living. The evidence seems to indicate that the introduction of MI to conventional treatment, with an adequate dose, may induce greater benefits over people with PD in early stages (I-III on the Hoehn and Yahr scale), especially in daily actions and movements functional such as gait, regardless of medication. However, the small sample size of the trials and the use of non-validated scales and non-objective tests, make it necessary that the results be viewed with caution. On the other hand, the cost-benefit ratio of the therapy, its benefits and its easy application are significant factors to take into account when adding MI to physiotherapy treatment in people with PD.

General objective: To determine whether gait training combined with MI exercises has a superior effect on gait, functionality in activities of daily living, motor capacity, and the perception of the quality of life in people with PD, which gait training without MI.

Specific objectives:

1. To study the validity of the instrumental technique available for the evaluation of gait and the intra- and inter-rater reliability with the same tool in healthy subjects.
2. To check the effect, in the short and medium-term, of a gait training program combined with MI in people diagnosed with PD.
3. To compare the effects of the gait and MI training program with the effects obtained through a gait rehabilitation program without MI exercises.
4. To contrast the gait pattern of people with PD before and after undergoing a rehabilitation program with MI, with that of healthy older people of the same age, sex, and height.
5. To observe the differences in the biomechanics of gait between the hemibody most affected by the signs of PD and the hemibody with less clinical alteration, before and after performing a gait training program combined with MI exercises.

Materials and Method:

The evaluation session will be carried out three times: before the treatment, at the end of the intervention, and 8-weeks after the intervention has finished. In each evaluation session, a clinical and biomechanical measurement will be carried out. The biomechanical evaluation will be done using 7 inertial sensors in a 10-meter walk corridor. The inertial sensor or inertial measurement unit (IMU) is made up of three different sensors: gyroscope, accelerometer, and magnetometer, capable of collecting information on the turns, linear acceleration, and magnetic north with respect to the earth's magnetic field. The part of the clinical evaluation includes the assessment of the functionality in the activities of daily living, the motor capacity, and the perception of the quality of life through different questionnaires and assessment scales.

Intervention:

Both, the experimental and control groups of this study, will perform an identical gait physiotherapy program, however, motor imagery exercises will be included in the experimental group.

The gait exercises are aimed at improving specific gait characteristics, so they will include:

* Exercises for length stride: walk with visual cues on the ground to reach a certain stride length, walk with horizontal poles at a height of 2 cm, walk over steps, treadmill walk.
* Exercises for Cadence training using a metronome.
* Exercises for gait velocity training by combining the visual and auditory feedback provided in previous exercises and on the treadmill
* Exercises for kinematic milestones during the stance and oscillation phase of gait through the mobility of the ankle, knee, and hip joints.

The motor imagery exercises will be performed in supine position on a stretcher, before each gait exercise. The instructions will be administered through the physiotherapy voice. The participant with closed eyes imagines himself performing the gait task while the general guidelines that guide the cognitive process are given. The instructions describe how the person is from the starting position and the different body movements that he must pay attention to during the imagining process. Through the instructions, the participant creates an image of himself and perceives the kinesthesia while performing the exercise. The duration of each motor imagery exercise is 8 minutes.

ELIGIBILITY:
The inclusion criteria are:

1. Diagnosed with PD according to the United Kingdom Parkinson's Disease Society Brain Bank diagnostic scale
2. Independent walk in a 10-meter corridor
3. Normal cognitive state, determined by the Mini-Mental State Examination with a score >25
4. Stable medication from the month before the start of the study until the t2 assessment.

Likewise, the exclusion criteria are:

1. Additional neurological condition different from PD
2. Disease or musculoskeletal acute alteration that limits mobility or balance
3. Lower extremities asymmetries >1 cm
4. Report pain on the Visual Analog Scale
5. Suffer from blindness, deafness, or any other visual/hearing impairment or pathology that may influence the ability to understand instructions and carry them out
6. Significant tremor that may interrupt the MI exercise
7. To perform other physical therapies or sports during the trial or the two months before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Gait velocity at the post-training time (primary time point) | 6 weeks
  Distance traveled by the body per unit of time at self-selected or comfortable speed, in the direction considered. It is expressed in meters per second (m / s).

SECONDARY OUTCOMES:
Gait speed variability | 6 weeks
  It is calculated through the coefficient of variation ([standard deviation/mean] × 100) of gait velocity. Indicates how stable or repeatable the participants are when walking.
Maximum gait speed | 6 weeks
  Distance traveled by the body per unit of time at the maximum possible speed, in the direction considered. It is expressed in meters per second (m/s).
Stance time | 6 weeks
  Time elapsed while the support or stance phase of the gait cycle is developed. It is expressed as a percentage of the total walking cycle and additionally in seconds.
Weight-acceptance Ground Reaction Force (Newton, N; Weight%) | 6 weeks
  Kinetic outcome; First force peak of vertical vector of the ground reaction forces during the stance phase of the gait cycle, which corresponds to the maximum reception of weight on the foot that initiates the gait cycle.
Midstance Ground Reaction Force (Newton, N; Weight%) | 6 weeks
  Kinetic outcome; Lowest force point of the valley located between both maximum force peaks of the vertical vector of the ground reaction forces, which corresponds to the swing of the opposite leg during the gait cycle.
Push-off Ground Reaction Force (Newton, N; Weight%) | 6 weeks
  Kinetic outcome; Second and last force peak of the vertical vector of the ground reaction forces during the stance phase of the gait cycle, which corresponds to the beginning of takeoff of the foot during the last part of the stance phase.
Breaking Ground Reaction Force (Newton, N; Weight%) | 6 weeks
  Kinetic outcome; First maximum force peak of the antero-posterior vector of the ground reaction forces during the gait cycle that corresponds to the braking of the foot on the ground.
Propulsion Ground Reaction Force (Newton, N; Weight%) | 6 weeks
  Kinetic outcome; Second maximum force peak of the antero-posterior vector of the ground reaction forces during the gait cycle that corresponds to the propulsion of the foot on the ground at the end of the stance phase.
Cadence (steps/min) | 6 weeks
  Number of steps executed in a time interval, its most commonly adopted unit being the step per minute.
Stride length | 6 weeks
  Distance measured between two consecutive supports points of the same foot; the heel strike is the reference used. It is expressed in meters (m).
Step length | 6 weeks
  The distance measured between one foot's heel contact and the other's heel contact. It is expressed in meters (m).
Swing time | 6 weeks
  Time elapsed while the swing phase develops. It is expressed as a percentage according to the entire walking cycle and additionally in seconds.
Double support time | 6 weeks
  Time that both feet are in contact with the ground during the gait cycle. It is expressed in seconds (s) and also as a percentage (%) of the total gait cycle.
Range of motion of lower limb joint (°) | 6 weeks
  Kinematic outcome that represents the range of motion in the sagittal plane of the hip, knee, and ankle joints performed during the gait cycle. These parameters will be specified for each limb (right and left).
Maximum ankle dorsiflexion during swing (°) | 6 weeks
  Kinematic outcome; Maximum ankle dorsiflexion angle reached during the swing phase, expressed in degrees.
Maximum knee flexion during swing (°) | 6 weeks
  Kinematic outcome; Maximum knee flexion angle reached during the swing phase, expressed in degrees.
Maximum hip extension during stance (°) | 6 weeks
  Kinematic outcome; Maximum hip extension angle reached during the stance phase, expressed in degrees.
Maximum hip flexion during swing (°) | 6 weeks
  Kinematic outcome; Maximum hip flexion angle reached during the swing phase, expressed in degrees.
Activities of daily life | 6 weeks
  Self-referred Quality of Life measured with the Schwab & England scale score.
Quality of Life perceived | 6 weeks
  Self-referred quality of life measured with the Parkinson's Disease Questionnaire-39 score questionnaire.
Freezing of gait | 6 weeks
  Freezing of gait Questionnaire score
Gait qualitative performance with TMT | 6 weeks
  Tinetti mobility test - Gait section score
Gait qualitative performance with DYPAGS | 6 weeks
  Dynamic Parkinson Gait Scale score
Balance qualitative performance with the TMT | 6 weeks
  Tinetti mobility test - Balance section score
Balance qualitative performance with the MiniBest | 6 weeks
  MiniBest test score
Mobility | 6 weeks
  Time taken to perform Timed-up and go test (s)

CONTACTS AND LOCATIONS:
Overall Officials: Constanza San Martín, PhD., Principal Investigator — Associate Lecturer professor at the Department of Physiotherapy
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
All measured and recorded data will be shared through the publications made and through their supplementary material.

REFERENCES:
- [Background] Leocadi M, Canu E, Sarasso E, Gardoni A, Basaia S, Calderaro D, Castelnovo V, Volonte MA, Filippi M, Agosta F. Dual-task gait training improves cognition and resting-state functional connectivity in Parkinson's disease with postural instability and gait disorders. J Neurol. 2024 Apr;271(4):2031-2041. doi: 10.1007/s00415-023-12151-w. Epub 2024 Jan 8. PMID 38189921
- [Background] Sarasso E, Gardoni A, Zenere L, Canu E, Basaia S, Pelosin E, Volonte MA, Filippi M, Agosta F. Action observation and motor imagery improve motor imagery abilities in patients with Parkinson's disease - A functional MRI study. Parkinsonism Relat Disord. 2023 Nov;116:105858. doi: 10.1016/j.parkreldis.2023.105858. Epub 2023 Sep 22. PMID 37774517
- [Background] Sarasso E, Agosta F, Piramide N, Gardoni A, Canu E, Leocadi M, Castelnovo V, Basaia S, Tettamanti A, Volonte MA, Filippi M. Action Observation and Motor Imagery Improve Dual Task in Parkinson's Disease: A Clinical/fMRI Study. Mov Disord. 2021 Nov;36(11):2569-2582. doi: 10.1002/mds.28717. Epub 2021 Jul 19. PMID 34286884
- [Background] Kashif M, Ahmad A, Bandpei MAM, Gilani SA, Hanif A, Iram H. Combined effects of virtual reality techniques and motor imagery on balance, motor function and activities of daily living in patients with Parkinson's disease: a randomized controlled trial. BMC Geriatr. 2022 Apr 30;22(1):381. doi: 10.1186/s12877-022-03035-1. PMID 35488213
- [Background] Kashif M, Ahmad A, Bandpei MAM, Gillani SA, Hanif A, Iram H. Effects of Virtual Reality with Motor Imagery Techniques in Patients with Parkinson's Disease: Study Protocol for a Randomized Controlled Trial. Neurodegener Dis. 2020;20(2-3):90-96. doi: 10.1159/000511916. Epub 2020 Dec 17. PMID 33333508
- [Background] Tinaz S, Kamel S, Aravala SS, Elfil M, Bayoumi A, Patel A, Scheinost D, Sinha R, Hampson M. Neurofeedback-guided kinesthetic motor imagery training in Parkinson's disease: Randomized trial. Neuroimage Clin. 2022;34:102980. doi: 10.1016/j.nicl.2022.102980. Epub 2022 Mar 2. PMID 35247729
- [Background] Santiago LM, de Oliveira DA, de Macedo Ferreira LG, de Brito Pinto HY, Spaniol AP, de Lucena Trigueiro LC, Ribeiro TS, de Sousa AV, Piemonte ME, Lindquist AR. Immediate effects of adding mental practice to physical practice on the gait of individuals with Parkinson's disease: Randomized clinical trial. NeuroRehabilitation. 2015;37(2):263-71. doi: 10.3233/NRE-151259. PMID 26484518
- [Background] Scarpina F, Magnani FG, Tagini S, Priano L, Mauro A, Sedda A. Mental representation of the body in action in Parkinson's disease. Exp Brain Res. 2019 Oct;237(10):2505-2521. doi: 10.1007/s00221-019-05608-w. Epub 2019 Jul 20. PMID 31327026
- [Background] Braun S, Beurskens A, Kleynen M, Schols J, Wade D. Rehabilitation with mental practice has similar effects on mobility as rehabilitation with relaxation in people with Parkinson's disease: a multicentre randomised trial. J Physiother. 2011;57(1):27-34. doi: 10.1016/S1836-9553(11)70004-2. PMID 21402327
- [Background] Bek J, Webb J, Gowen E, Vogt S, Crawford TJ, Sullivan MS, Poliakoff E. Patients' Views on a Combined Action Observation and Motor Imagery Intervention for Parkinson's Disease. Parkinsons Dis. 2016;2016:7047910. doi: 10.1155/2016/7047910. Epub 2016 Sep 29. PMID 27777809
- [Background] Bek J, Gowen E, Vogt S, Crawford TJ, Poliakoff E. Combined action observation and motor imagery influences hand movement amplitude in Parkinson's disease. Parkinsonism Relat Disord. 2019 Apr;61:126-131. doi: 10.1016/j.parkreldis.2018.11.001. Epub 2018 Nov 9. No abstract available. PMID 30470657
- [Background] Subramanian L, Morris MB, Brosnan M, Turner DL, Morris HR, Linden DE. Functional Magnetic Resonance Imaging Neurofeedback-guided Motor Imagery Training and Motor Training for Parkinson's Disease: Randomized Trial. Front Behav Neurosci. 2016 Jun 8;10:111. doi: 10.3389/fnbeh.2016.00111. eCollection 2016. PMID 27375451
- [Background] Bezerra PT, Santiago LM, Silva IA, Souza AA, Pegado CL, Damascena CM, Ribeiro TS, Lindquist AR. Action observation and motor imagery have no effect on balance and freezing of gait in Parkinson's disease: a randomized controlled trial. Eur J Phys Rehabil Med. 2022 Oct;58(5):715-722. doi: 10.23736/S1973-9087.22.07313-0. Epub 2022 Sep 1. PMID 36052889
- [Background] Tamir R, Dickstein R, Huberman M. Integration of motor imagery and physical practice in group treatment applied to subjects with Parkinson's disease. Neurorehabil Neural Repair. 2007 Jan-Feb;21(1):68-75. doi: 10.1177/1545968306292608. PMID 17172556